CLINICAL TRIAL: NCT05534919
Title: An Open-label Extention (OLE) Study to Evaluate the Efficacy and Safety of Nefecon Treatment in Patients with IgA Nephropathy Who Have Completed Study Nef-301 in China
Brief Title: Efficacy and Safety in Chinese Patients with Immunoglobulin a Nephropathy (IgAN) Who Have Completed Study Nef-301
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Everest Medicines (Singapore) Pte. Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ES103002
Record Dates: First submitted 2022-09-06; First posted 2022-09-10 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-01

CONDITIONS: Primary Immunoglobulin a Nephropathy (IgAN)
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Intervention Model Description: This is an open label, single-arm study with active treatment.
Masking Description: This is an open label, single-arm study with active treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nefecon active treatment (Experimental): Nefecon 16mg once daily for 9 months.
  Interventions: Drug: Nefecon

INTERVENTIONS:
Drug: Nefecon — Nefecon is taken orally as capsules once daily for 9 months.

SUMMARY:
This is a Phase 3b, multicenter, open-label extension (OLE) study to evaluate the efficacy and safety of Nefecon treatment in Chinese patients who have completed Nef-301 and continue to be treated with a stable dose of Renin-angiotensin system (RAS) inhibitor therapy (Angiotensin-converting enzyme inhibitors (ACEIs) and/or Angiotensin II type I receptor blockers (ARBs).

DETAILED DESCRIPTION:
This is a Phase 3b, multicenter, open-label extension (OLE) study to evaluate the efficacy and safety of Nefecon treatment in Chinese patients with Immunoglobulin A nephropathy (IgAN) who have completed Nef 301 study and continue to be treated with a stable dose of RAS inhibitor therapy (ACEIs and/or ARBs).

During Study open-label extension (OLE) study, patients will receive Nefecon for a 9-month period. The patient will come for a follow-up visit at 12 months after first dose.

ELIGIBILITY:
Inclusion Criteria:

1. Patients that completed study Nef-301.
2. On a stable dose of RAS inhibitor therapy (ACEIs and/or ARBs) at the maximum allowed dose or maximum tolerated dose according to the 2012 Kidney Disease: Improving Global Outcomes (KDIGO) guidelines.
3. Willing and able to provide written informed consent.
4. Urine protein to creatinine ratio (UPCR) equal to or more than 0.5 g/gram or Average proteinuria equal or more than 0.75 g/day.
5. eGFR equal to or more than 30 mL/min per 1.73 m2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula.

Exclusion Criteria:

1. Systemic diseases that may cause mesangial Immunoglobulin A (IgA) deposition.
2. Patients who have undergone a kidney transplant.
3. Patients with presence of other glomerulopathies and/or nephrotic syndrome.
4. Patients with acute, chronic, or latent infectious disease including hepatitis, tuberculosis (TB), human immunodeficiency virus (HIV), and chronic urinary tract infections.
5. Patients with liver cirrhosis, as assessed by the Investigator.
6. Patients with a diagnosis of type 1 or type 2 diabetes mellitus which is poorly controlled.
7. Patients with history of unstable angina, class III or IV congestive heart failure, and/or clinically significant arrhythmia, as judged by the Investigator.
8. Patients with unacceptable blood pressure control defined as a blood pressure consistently above national guidelines for proteinuric renal disease, as assessed by the Investigator.
9. Patients with diagnosed malignancy within the past 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Change in urine protein to creatinine ratio (UPCR) after 9 months | 9 months
  The outcome is measured as urine protein to creatinine ratio (UPCR) based on 24 hour urine collections at 9 months following the first dose of Nefecon compared to baseline.following the first dose of Nefecon compared to baseline.
Change in estimated glomerular filtration rate(eGFR) at 9 months | 9 months
  The outcome is measured as change in eGFR at 9 months following the first dose of Nefecon compared to baseline.
The incidence of treatment emergent adverse events | from enrollment up to 12 months
  Adverse event data collection

CONTACTS AND LOCATIONS:
Overall Officials: Jicheng Lv, Doctor, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No